CLINICAL TRIAL: NCT05128630
Title: An Open-label, Multi-center, Phase 2 Study of Chemo-immunotherapy Followed by Reduced-dose Hypo-fractionated RT and Maintenance Immunotherapy for Stage III Unresectable Non -Small-cell Lung Carcinoma (NSCLC).
Brief Title: Chemo-immunotherapy, Hypo-fractionated RT and Maintenance Immunotherapy for Stage III NSCLC.
Acronym: DEDALUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Andrea Riccardo Filippi, prof., Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210040686
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: NSCLC, Stage III
Keywords: durvalumab; radiotherapy; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: open-label, multi-center, single arm phase 2 trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm (Experimental): Chemotherapy plus durvalumab, hypofractionated RT plus durvalumab, durvalumab maintenance
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Patients will receive 1500 mg durvalumab via IV infusion q3w concomitant with chemotherapy (Cisplatin/carboplatin plus etoposide) for up to a maximum of 3 cycles, then via IV infusion at the same interval during sequential radiotherapy and then every 4 weeks for up to a maximum of 12 months or until confirmed disease progression, unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.
  Other Names: radotherapy; chemotherapy

SUMMARY:
Aim of this phase 2 study is to evaluate the safety and the efficacy of the combination of induction chemotherapy plus durvalumab followed by reduced-dose hypo-fractionated thoracic RT (concurrent with durvalumab) and durvalumab maintenance for stage 3 unresectable NSCLC patients candidate to sequential chemo-RT.

DETAILED DESCRIPTION:
The study hypothesis is that the new regimen tested in this study will be safe and effective by:

1. anticipating the use of durvalumab, together with chemotherapy (higher efficacy)
2. harnessing response to induction chemo-durvalumab (which is expected to be significant) to be able to reduce radiotherapy dose without reducing tumor control probability
3. reducing radiation-induced immunosuppression
4. reducing radiation-induced late morbidity, this aspect is important when considering that this regimen is expected to be able to cure a proportion of patients (long-term survivors)

In this phase II study, the investigators will evaluate the combination of induction chemotherapy plus durvalumab followed by reduced-dose hypo-fractionated thoracic RT (concurrent with durvalumab) and durvalumab maintenance for stage 3 unresectable NSCLC patients candidate to sequential chemo-RT.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
2. Provision of signed and dated, written ICF prior to any mandatory study specific procedures, sampling, and analyses.

   Age
3. 18 years or older at the time of signing the ICF. Type of patient and disease characteristics
4. Histologically- or cytologically-documented NSCLC with locally-advanced, unresectable Stage III disease (according to the IASLC Staging Manual Version 8 [IASLC 2016]). Positron emission tomography (PET)/CT, MRI of the brain, and endobronchial ultrasound with biopsy are highly encouraged at diagnosis.
5. Patients with measurable disease assessed at baseline by CT/MRI will be entered in this study.
6. Must have a life expectancy of at least 12 weeks at enrolment.
7. WHO/ECOG PS 0-1.
8. Patient not eligible for concurrent chemo radiation according to investigator assessment
9. Adequate organ and marrow function at enrollment as defined below. These parameters should be achieved without augmentation by growth factors, transfusions, or infusions within 28 days of screening unless required for SoC:

   1. Haemoglobin ≥9.0 g/dL;
   2. Absolute neutrophil count >1.0 × 109/L;
   3. Platelet count >75 × 109/L;
   4. Serum bilirubin ≤1.5 × upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed in consultation with their physician.
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN.
   6. Measured creatinine clearance >40 mL/min or calculated creatinine clearance >40 mL/min as determined by Cockcroft-Gault (using actual body weight) (Cockcroft and Gault 1976).

   Males:

   Creatinine clearance (mL/min) = [Weight (kg) × (140 - Age)] / 72 × serum creatinine (mg/dL)

   Females:

   Creatinine clearance (mL/min) = [Weight (kg) × (140 - Age) × 0.85] / 72 × serum creatinine (mg/dL)
10. Body weight >30 kg at enrollment
11. Male or female. Reproduction
12. Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    1. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).

Exclusion Criteria:Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Patients who have disease considered for surgical treatment as part of their care plan, such as Pancoast or superior sulcus tumors.
2. Mixed small-cell lung cancer and NSCLC histology.
3. History of allogeneic organ transplantation.
4. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia.
   2. Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement.
   3. Any chronic skin condition that does not require systemic therapy.
   4. Patients without active disease in the last 5 years at enrolment may be included but only after consultation with the Study Physician.
   5. Patients with celiac disease controlled by diet alone.
5. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, ILD, serious chronic GI conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
6. History of another primary malignancy except for:

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. Adequately treated carcinoma in situ without evidence of disease.
7. History of leptomeningeal carcinomatosis.
8. History of active primary immunodeficiency.
9. Active infection including hepatitis B (known positive hepatitis B surface antigen [HbsAg] result), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies). Patients with a past or resolved hepatitis B virus (HBV) infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HbsAg) are eligible. Patients positive for hepatitis C antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
10. Any unresolved toxicity of NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

    1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
    2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
11. Known allergy or hypersensitivity to durvalumab or any of the IP excipients. Prior/concomitant therapy
12. Prior chemo-radiotherapy for lung cancer. Prior surgical resection (ie, Stage I or II) is permitted.
13. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.

    Note: Patients, if enrolled, should not receive live vaccine while receiving IP and up to 30 days after the last dose of IP.
14. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.

Note: Local surgery of isolated lesions for palliative intent is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-11-28 (Estimated); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Safety | Within 6 months from study enrollment
  Incidence of Grade 3 or more possibly related adverse events (PRAEs)

SECONDARY OUTCOMES:
Progression-Free Survival | 0-36 months from study enrollment
  Kaplan-Meier Progression-Free Survival, according to RECIST 1.1 and as assessed by the Investigators
Overall Survival | 0-36 months from study enrollment
  Kaplan-Meier Overall Survival

OTHER OUTCOMES:
Quality of Life | 0-36 months
  EORTC QLQ-C30 and LC13

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No